CLINICAL TRIAL: NCT02176018
Title: A Randomized Pilot Study of Nuedexta for the Prevention and Modification of Disease Progression in Episodic Migraine
Brief Title: Nuedexta for the Prevention and Modification of Disease Progression in Episodic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-001AV
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Episodic Migraine
Keywords: Episodic Migraine; Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nuedexta (Active Comparator): One capsule will be taken (dextromethorphan HB and quinidine sulfate, 20 mg/10 mg) daily for seven days. On the eight day and for the remainder of the study 2 capsule will be taken twice a day. Medication will be taking daily for a total of 3 months.
  Interventions: Drug: Dextromethorphan and quinidine
- Placebo (Placebo Comparator): One capsule will be taken of placebo to match daily for seven days. On the eight day and for the remainder of the study 2 capsule will be taken twice a day. Medication will be taking daily for a total of 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan and quinidine
  Other Names: Nuedexta
  Arms: Nuedexta
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and effectiveness of daily dextromethorphan/quinidine (Nuedexta) in reducing the frequency and progression of episodic migraine.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, multi-center study to be conducted at the Headache Care Center in Springfield, MO and two other clinics in the United States. Approximately 45 subjects, 18 to 65 years of age, with frequent episodic migraine (6-14 days per month), with (1.2) or without aura (1.1) as defined by ICHD-3beta, will enter a 1-month baseline period to confirm the migraine diagnosis, as well as establish baseline characteristics. At Visit 1, subjects must not have a history of utilization of acute treatment greater than 14 days per month in the preceding 3 month period. Subjects must have a current history of ICHD-3beta migraine with 6-14 migraine days per month in the 3 months prior to the study enrollment. Eligible subjects will be randomly assigned to one of two groups in a 1:1 ratio. Randomization will occur using a computer-generated allocation schedule. Subjects meeting entrance criteria as determined both at screening and through the review of the baseline headache diary will be given the lowest available allocation number for that site. Migraine preventative use is permitted if the subject has been on a stable does for at least 2 months prior to screening and has not failed more than 3 migraine preventatives due to lack of efficacy. The study will consist of 5 office visits per subject: Visit 1 - screening, Visit 2 - randomization, and Visits 3 to 5 - three-month treatment period. During the baseline period, the subject will treat migraines with their current preferred acute treatment of choice.

ELIGIBILITY:
Inclusion Criteria:

* male or female, in otherwise good health, 18 to 65 years of age.
* history of frequent episodic migraine for at least 3 months as defined by 6-14 migraine days per month with or without aura according to the ICHD-3beta or a migraine treated with an ergot or triptan which resulted in relief.
* onset of migraine before age 50.
* stable history of headache at least 3 months prior to screening.
* if using daily migraine preventive medications for migraine or for other medical conditions (e.g. propranolol being used for hypertension) and has been on a stable dose and regimen for at least 2 months prior to beginning the baseline period.
* female, of childbearing potential, and agrees to maintain true abstinence or use (or have their partner use) one of the listed methods of birth control for the duration of the study: hormonal contraceptive, intrauterine device (IUD), condoms, diaphragm, and/or vasectomy. The use of barrier contraceptive (condom or diaphragm) should always be supplemented with the use of a spermicide. Note: To be considered not of childbearing potential, subject must be 6 weeks post-surgical bilateral oophorectomy, hysterectomy, or bilateral tubal ligation, or postmenopausal for at least one year.

Exclusion Criteria:

* unable to understand the study requirements, the informed consent, or complete headache records as required per protocol.
* pregnant, actively trying to become pregnant, or breast-feeding.
* female of childbearing potential not using adequate contraceptive measures.
* experienced the following migraine variants: basilar migraine, aura without headache, familial hemiplegic migraine, complicated migraine, ophthalmoplegic migraine and retinal migraine.
* history of Medication Overuse Headache (Appendix II) in the 3 months prior to study enrollment or during the baseline phase.
* history of acute migraine treatment greater than 14 days per month in 3 months prior to screening.
* history of 3 or more failed preventative medications due to lack of efficacy for prophylactic treatment of migraine after an adequate therapeutic trial.
* received onabotulinumtoxinA injections within 3 months prior to screening and/or will receive onabotulinumtoxinA injections during the study.
* abused, in the opinion of the Investigator, any of the following drugs, currently or within the past 1 year: opioids, alcohol, barbiturates, benzodiazepine, cocaine.
* taken, or plans to take: a monoamine oxidase inhibitor (MAOI) including herbal preparations containing St. John's wort (Hypericum perforatum) within 14 days of Visit 1, concomitant medications and/or foods containing dextromethorphan, quinidine, quinine, mefloquine, paxil, dicyclomine, digitalis, thioridazine or pimozide (medications that prolong QT interval) anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
* history of hypersensitivity to medications containing dextromethorphan.
* history of hypersensitivity to medications or foods containing quinidine.
* at an increased risk of developing serotonin syndrome, in the opinion of the investigator.
* history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study.
* unstable neurological condition or a significantly abnormal neurological examination with focal signs or signs of increased intracranial pressure.
* cardiovascular disease (ischemic heart disease, including angina pectoris, myocardial infarction, documented silent ischemia, or with Prinzmetal's angina); has symptoms of ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome.
* ECG results outside normal limits (> 470 msec), prolonged QT interval, congenital long QT syndrome, torsades de pointes, or complete AV block.
* has uncontrolled hypertension (≥ 140/90mmHg in either the systolic or diastolic measurements in 2 out of 3 BP readings at screening).
* serious illness, or an unstable medical condition, one that could require hospitalization, or could increase the risk of adverse events, in the opinion of the investigator.
* any psychiatric disorder with psychotic features and any other psychiatric disorder not stable or well controlled, that would interfere in their ability to complete study activities.
* received any investigational agents within 30 days prior to Visit 1.
* plans to participate in another clinical study at any time during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Swedish American Neuro and Headache Center, Rockford, Illinois
  - The Headache Center, Ridgeland, Mississippi
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Clinvest, Springfield, Missouri
  - Island Neurological Associates, PC, Plainview, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 90 participants were screened, 14 failed to meet the inclusion criteria and were screen failed. 76 participants were enrolled into a 28-day run-in period. 31 were excluded from the study prior to being assigned to a treatment arm, due to failure to meet inclusion criteria. A total of 45 participants were randomized.
Groups:
- Nuedexta: One capsule will be taken (dextromethorphan HB and quinidine sulfate, 20 mg/10 mg) daily for seven days. On the eight day and for the remainder of the study 2 capsule will be taken twice a day. Medication will be taking daily for a total of 3 months.
  Dextromethorphan and quinidine
- Placebo: One capsule will be taken of placebo to match daily for seven days. On the eight day and for the remainder of the study 2 capsule will be taken twice a day. Medication will be taking daily for a total of 3 months.
  Placebo
Period: Overall Study
Arm/Group | Nuedexta | Placebo
Started | 22 | 23
Completed | 17 | 17
Not Completed | 5 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nuedexta | Placebo | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.23 (9.62) | 44.17 (11.62) | 44.69 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 23 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45
Headache Days [Mean (Standard Deviation); unit: Number of Headache Days] — Number of headache days reported during the 28 day run-in period. Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. These criteria excluded 6 subjects in the Placebo arm and 2 subjects in the Nuedexta arm from the analysis data sets. Thus, 37 participants were analyzed for this Baseline Measurement.
  Number of Headache Days
    number analyzed (Participants) | 20 | 17 | 37
    (all) | 10.5 (2.5) | 10.29 (5.28) | 10.4 (3.96)
Migraine Days [Mean (Standard Deviation); unit: Number of Migraine days] — Number of migraine days reported during the 28 day run-in period. Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. These criteria excluded 6 subjects in the Placebo arm and 2 subjects in the Nuedexta arm from the analysis data sets. Thus, 37 participants were analyzed for this Baseline Measurement.
  Number of Migraine days
    number analyzed (Participants) | 20 | 17 | 37
    (all) | 9 (2.15) | 8 (2.5) | 8.54 (2.34)
Headache Severity [Mean (Standard Deviation); unit: units on a scale] — Headache pain severity reported during the 28 day run-in period. Measured on a scale from 1 = Mild, to 3 = Severe. Higher numbers indicating more severe headache pain. Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. These criteria excluded 6 subjects in the Placebo arm and 2 subjects in the Nuedexta arm from the analysis data sets. Thus, 37 participants were analyzed for this Baseline Measurement.
  units on a scale
    number analyzed (Participants) | 20 | 17 | 37
    (all) | 2.02 (0.386) | 2.17 (0.326) | 2.09 (0.362)
Headache Duration [Mean (Standard Deviation); unit: Hours] — Average headache duration reported during the 28 day run-in period, measured in hours. Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. These criteria excluded 6 subjects in the Placebo arm and 2 subjects in the Nuedexta arm from the analysis data sets. Thus, 37 participants were analyzed for this Baseline Measurement.
  Hours
    number analyzed (Participants) | 20 | 17 | 37
    (all) | 6.14 (2.12) | 5.54 (2.03) | 5.86 (2.07)
Acute Medication Use [Mean (Standard Deviation); unit: Number of medications] — Number of doses of acute medication taken, reported during the 28 day run-in period. Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. These criteria excluded 6 subjects in the Placebo arm and 2 subjects in the Nuedexta arm from the analysis data sets. Thus, 37 participants were analyzed for this Baseline Measurement.
  Number of medications
    number analyzed (Participants) | 20 | 17 | 37
    (all) | 16.4 (9.58) | 13.4 (7.44) | 15.0 (8.68)

OUTCOME MEASURES:

1. Primary Outcome: Headache Days in Each Treatment Period Month
Description: The average number of headache days at treatment period months 1, 2, and 3 (28 day periods for each month) for the Nuedexta arm and the Placebo arm. Headache days were defined as any patient reported head pain during the prior 24 hour period.
Time Frame: Treatment Month 1, Treatment Month 2, and End of Treatment Period Month 3 (Day 116)
Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. These criteria excluded 6 subjects in the Placebo arm and 2 subjects in the Nuedexta arm from the analysis data sets. Thus, 37 participants were analyzed for this measure.
Measure: Mean (Standard Deviation); unit: Number of Headache days
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 20 | 17
Number of Headache days
  Treatment Month 1 | 7.1 (3.31) | 10.88 (6.25)
  Treatment Month 2 | 7.05 (3.82) | 9.47 (6.15)
  Treatment Month 3 | 7.10 (3.8) | 9.77 (7.09)

2. Secondary Outcome: Headache Days in Treatment Period Month 3
Description: The average number of headache days at treatment period month 3 (28 day period) for the Nuedexta arm and the Placebo arm. Headache days were defined as any patient reported head pain during the prior 24 hour period.
Time Frame: End of Treatment Period Month 3 (Day 116)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of headache days
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 20 | 17
Number of headache days | 7.1 (3.8) | 9.77 (7.09)

3. Secondary Outcome: Migraine Days in Each Treatment Period Month
Description: The average number of migraine days at treatment period months 1, 2, and 3 (28 day periods for each month) for the Nuedexta arm and the Placebo arm.
Time Frame: Treatment Month 1, Month 2, and End of Treatment Period Month 3 (Day 116)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Migraine days
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 20 | 17
Number of Migraine days
  Treatment Month 1 | 5.65 (3.35) | 7.65 (2.71)
  Treatment Month 2 | 5.85 (3.48) | 6.94 (4.05)
  Treatment Month 3 | 6.05 (3.63) | 7.29 (4.3)

4. Secondary Outcome: Headache Severity in Each Treatment Period Month
Description: The average headache severity at treatment period months 1, 2, and 3 (28 day periods for each month) for the Nuedexta arm and the Placebo arm. Headache pain severity was measured on a scale from 1 = Mild, to 3 = Severe. Higher numbers indicating more severe headache pain.
Time Frame: Treatment Month 1, Month 2, and End of Treatment Period Month 3 (Day 116)
Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. Additionally, participants who were unavailable for the assessment at a particular time point were excluded. These criteria excluded 6 subjects in the Placebo arm and 3 subjects in the Nuedexta arm from the analysis data sets.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 19 | 17
units on a scale
  Treatment Month 1 | 1.69 (0.37) | 2.04 (0.43)
  Treatment Month 2 | 1.81 (0.52) | 1.96 (0.45)
  Treatment Month 3 | 1.74 (0.46) | 1.86 (0.51)

5. Secondary Outcome: Headache Duration in Each Treatment Period Month
Description: The average headache duration (time of onset to pain free) at treatment period months 1, 2, and 3 (28 day periods for each month) for the Nuedexta arm and the Placebo arm. Headache duration was measured in hours.
Time Frame: Treatment Month 1, Month 2, and End of Treatment Period Month 3 (Day 116)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 19 | 17
Hours
  Treatment Month 1 | 5.39 (2.38) | 5.30 (2.25)
  Treatment Month 2 | 6.33 (4.06) | 5.75 (2.78)
  Treatment Month 3 | 6.60 (4.81) | 5.46 (2.72)

6. Secondary Outcome: 50% Headache Reduction
Description: The number of subjects with at least a 50% reduction in number of headache days comparing baseline to each visit (treatment period months 1, 2, and 3: 28 day for each month) in the Nuedexta arm vs. the placebo arm.
Time Frame: Baseline (Day 0) to Treatment Period Month 3 (Day 116)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 20 | 17
Participants
  Treatment Month 1 | 6 | 0
  Treatment Month 2 | 7 | 2
  Treatment Month 3 | 8 | 8

7. Secondary Outcome: Acute Medication Use in Each Treatment Period Month
Description: The average number of doses of acute medication taken at treatment period months 1, 2, and 3 (28 day periods for each month) for the Nuedexta arm and the Placebo arm
Time Frame: Treatment Month 1, Month 2, and End of Treatment Period Month 3 (Day 116)
Population: Randomized subjects were required to complete at least one full month of treatment period to be included in the analyses. These criteria excluded 6 subjects in the Placebo arm and 2 subjects in the Nuedexta arm from the analysis data sets.
Measure: Mean (Standard Deviation); unit: Number of medication doses
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 20 | 17
Number of medication doses
  Treatment Month 1 | 9.45 (6.82) | 13.06 (12.30)
  Treatment Month 2 | 9.50 (7.08) | 11.41 (12.52)
  Treatment Month 3 | 11.55 (11.01) | 10.94 (12.95)

8. Secondary Outcome: Migraine Disability Assessment Scale (MIDAS)
Description: MIDAS scores at Visit 2 and Visit 5 (end of treatment period month 3). The MIDAS is a questionnaire consisting of five (5) "how many days in the last 3 months..." questions. Thus the range for the MIDAS is from, 0 to a maximum possible score 93 (31 days X 3 months). The MIDAS is scored according to the following:
  0-5, MIDAS Grade I, Little or No Disability 6-10, MIDAS Grade II, Mild Disability 11-20, MIDAS Grade III, Moderate Disability 21+, MIDAS Grade IV, Severe Disability
Time Frame: Visit 2 (Day 28) to Visit 5 (Day 116)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Visit 2 (Day28) | 34.95 (22.65) | 32.88 (29.95)
  Visit 5 (Day 116) | 22.50 (17.41) | 30.35 (42.47)

9. Secondary Outcome: Headache Health Score
Description: Headache Health Score at Visit 2 (Day 28), Visit 3 (Day 57), Visit 4 (Day 85), and Visit 5 (Day 116) for the Nuedexta arm and the placebo arm. The Headache Health Score is measured using a scale from 0 to 100, with higher scores indicating less headache impact on the subject's life.
Time Frame: Visit 2 (Day 28), Visit 3 (Day 57), Visit 4 (Day 85), and Visit 5 (Day 116)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Visit 2 (Day 28) | 78.71 (5.25) | 81.07 (7.37)
  Visit 3 (Day 57) | 87.62 (6.57) | 80.30 (10.62)
  Visit 4 (Day 85) | 87.14 (8.31) | 82.28 (10.77)
  Visit 5 (Day 116) | 87.57 (6.97) | 84.10 (10.76)

10. Secondary Outcome: Adverse Events
Description: Compare the number of adverse events in the Nuedexta arm vs. the placebo arm.
Time Frame: Baseline (Day 0) to Treatment Period Month 3 (Day 116)
Measure: Number; unit: Number of Adverse Events
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 22 | 23
Number of Adverse Events | 9 | 35

ADVERSE EVENTS:
Time Frame: 116 days
Arm/Group | Nuedexta | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/23
Other Adverse Events (participants affected / at risk) | 4/22 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nuedexta (N=22) | Placebo (N=23)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nuedexta (N=22) | Placebo (N=23)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 1 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02176018/SAP_000.pdf
  • Study Protocol (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02176018/Prot_001.pdf